CLINICAL TRIAL: NCT02092805
Title: Repetitive Transcranial Magnetic Stimulation in Visceral Pain Secondary to Malignancy
Brief Title: rTMS as a Treatment of Visceral Pain Secondary to Malignancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Eman M. Khedr, Clinical rofessor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: rTMS in malig. visceral pain
Record Dates: First submitted 2014-03-19; First posted 2014-03-20 (Estimated); Last update posted 2014-03-20 (Estimated); Status verified 2014-03

CONDITIONS: Malignancy
Keywords: VAS; VDS; HAM-D; Visceral pain; Malignancy; rTMS; Motor cortex; Analgesia; Dynorphin
MeSH Terms: conditions — Neoplasms; Visceral Pain; Agnosia; Spinocerebellar ataxia 23

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sham rTMS (Sham Comparator): Sham-rTMS was applied using the same parameters but with the coil elevated and angled away from the head to reproduce some of subjective sensation of rTMS.
  Interventions: Procedure: Sham rTMS (same parameters but with coil elevated and angled away from the head) every day for 10 consecutive days (5 days/week).
- Real rTMS (Active Comparator): The active group recieved real-rTMS over the motor cortical area corresponding to the hand of painful side. Each train consist of 2000 pulses at 20 Hz and 80% RMT (total duration 10s). The treatment was repeated every day for 5 consecutive days in week for two weeks (the total number of sessions had be given was 10 sessions).
  Interventions: Procedure: Real rTMS(20 Hz, 10 trains, inter train interval 30 sc with total pulses 2000, intensity 80% of motor threshold) daily for 10 consecutive days (5 days/week)

INTERVENTIONS:
Procedure: Real rTMS(20 Hz, 10 trains, inter train interval 30 sc with total pulses 2000, intensity 80% of motor threshold) daily for 10 consecutive days (5 days/week)
  Arms: Real rTMS
Procedure: Sham rTMS (same parameters but with coil elevated and angled away from the head) every day for 10 consecutive days (5 days/week).
  Arms: Sham rTMS

SUMMARY:
The purpose of this study is to assess the efficacy of rTMS over primary motor cortex in patients suffering from malignant visceral pain. Thirty four patients were included in the study. They are divided randomly into 2 groups using closed envelop as real rTMS group and sham group. Real rTMS over the hand area of motor cortex (20 Hz, 10 trains with inter train interval 30 second with total pulses 2000, intensity 80% of motor threshold) every day for ten consecutive days (5 days/week) and the coil elevated and angled away from the head as sham stimulation. Patients were evaluated by verbal descriptor scale (VDS), visual analog scale (VAS), and Hamilton rating scale for depression (HAM-D) at the baseline, after 1st, 5th, 10th session, 15 day and 1 month after end of sessions. Serum human dynorphin (Dyn) level was measured at baseline, 5th and 10th session.

ELIGIBILITY:
Inclusion Criteria:

* All patients within age group 18-65 years with malignant visceral pain resistant to medical treatment for at least 2 months or associated with significant adverse effect from medication was involved in this study.

Exclusion Criteria:

* We excluded patients with intracranial metallic devices or with pacemakers or any other device. We also excluded those with extensive myocardial ischemia, unstable angina and those known to have epilepsy.

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2010-01; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Visceral pain improvement | one month
  Reduction of visceral pain in patients with malignancy measured by VAS, VDS.

SECONDARY OUTCOMES:
Reduction of depression manifestation | one month
  Measurement of depression by using (HAM-D) scale.